CLINICAL TRIAL: NCT00719667
Title: German Off Pump Coronary Artery Bypass in Elderly Study
Acronym: GOPCABE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German Off Pump Coronary Artery Bypass in Elderly Study Group (Network)
Collaborators: Institut für Klinisch-Kardiovaskuläre Forschung GmbH (Network); Deutsche Gesellschaft für Herz-, Thorax- und Gefäßchirurgie (Unknown)
Responsible Party: Principal Investigator, PD Dr. Michael Hilker, Professor Hilker, German Off Pump Coronary Artery Bypass in Elderly Study Group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: op 001
Record Dates: First submitted 2008-07-20; First posted 2008-07-22 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Heart Disease
Keywords: OPCAB; coronary; bypass; grafting; off pump
MeSH Terms: conditions — Heart Diseases | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: coronary artery bypass grafting — on pump off pump

SUMMARY:
Comparison of two operative techniques (on-pump vs off-pump)of coronary revascularisation of the best treatment concept for patients older or 75 years old.

Hypothesis: The coronary bypass operation without use of the heart-lung machine (off-pump=OPCAB) reduces the combined endpoint in comparison with the conventional coronary bypass operation (on-pump).

ELIGIBILITY:
Inclusion Criteria:

* older or 75 years
* indication for elective bypass operation
* patient has signed written consent before randomization

Exclusion Criteria:

* previous heart surgery
* patient unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 1 month and 12 month
Myocardial infarction | 1 month and 12 month
Stroke | 1 month and 12 month
Any revascularisation | 1 month and30 month
renal failure | 1 month and 12 month

SECONDARY OUTCOMES:
ventilation time | post op
blood transfusion | post op
length of stay in intensive-care unit | post op

CONTACTS AND LOCATIONS:
Overall Officials: Anno Diegeler, Professor, Principal Investigator — Herzchirurgie Bad Neustadt/Saale; Michael Hilker, PD, Study Chair — Universität Regensburg
Locations (2):
- Germany (2):
  - Herzchirurgie Neustadt/Saale, Neustadt/Saale, Bavaria
  - Universität Regensburg, Regensburg, Bavaria

REFERENCES:
- [Derived] Diegeler A, Borgermann J, Kappert U, Hilker M, Doenst T, Boning A, Albert M, Farber G, Holzhey D, Conradi L, Riess FC, Veeckmann P, Minorics C, Zacher M, Reents W. Five-Year Outcome After Off-Pump or On-Pump Coronary Artery Bypass Grafting in Elderly Patients. Circulation. 2019 Apr 16;139(16):1865-1871. doi: 10.1161/CIRCULATIONAHA.118.035857. PMID 30732456
- [Derived] Faerber G, Zacher M, Reents W, Boergermann J, Kappert U, Boening A, Diegeler A, Doenst T; GOPCABE investigators. Female sex is not a risk factor for post procedural mortality in coronary bypass surgery in the elderly: A secondary analysis of the GOPCABE trial. PLoS One. 2017 Aug 30;12(8):e0184038. doi: 10.1371/journal.pone.0184038. eCollection 2017. PMID 28854266
- [Derived] Diegeler A, Borgermann J, Kappert U, Breuer M, Boning A, Ursulescu A, Rastan A, Holzhey D, Treede H, Riess FC, Veeckmann P, Asfoor A, Reents W, Zacher M, Hilker M; GOPCABE Study Group. Off-pump versus on-pump coronary-artery bypass grafting in elderly patients. N Engl J Med. 2013 Mar 28;368(13):1189-98. doi: 10.1056/NEJMoa1211666. Epub 2013 Mar 11. PMID 23477657